CLINICAL TRIAL: NCT04426981
Title: Behavioral Activation in Orthopaedic Trauma Patients: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D20133
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Fractures, Bone
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Consenting patients will be enrolled into a Behavioral Activation treatment arm. Behavioral activation is a behavioral treatment that focuses on helping participants engage in more rewarding and enjoyable activities.
  Interventions: Behavioral: Behavioral Activation

INTERVENTIONS:
Behavioral: Behavioral Activation — Behavioral activation is a behavioral treatment that focuses on helping participants engage in more rewarding and enjoyable activities. In the first session, participants will begin to identify domains of their life which are important to them. In the second session, participants will be assisted in creating an action plan to engage in more activities in one or more domains of importance. In session 3-8, participants will be assisted in problem solving any challenges they encountered in implementing their previous action plan and will develop a new action plan. The intervention will continue until participants achieved three action plans or reach the eight-session limit, whichever comes first.

SUMMARY:
This is a prospective observational pilot study designed to evaluate feasibility and acceptability as well as preliminary efficacy of a behavioral activation intervention among orthopaedic trauma patients after discharge home following their injury.

DETAILED DESCRIPTION:
This is a prospective observational pilot study designed to evaluate feasibility and acceptability as well as preliminary efficacy of a behavioral activation intervention among orthopaedic trauma patients after discharge home following their injury. Behavioral activation is a behavioral treatment that focuses on helping participants engage in more rewarding and enjoyable activities. In the first session, participants will begin to identify domains of their life which are important to them. In the second session, participants will be assisted in creating an action plan to engage in more activities in one or more domains of importance. In session 3-8, participants will be assisted in problem solving any challenges they encountered in implementing their previous action plan and will develop a new action plan. The intervention will continue until participants achieved three action plans or reach the eight-session limit, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Presenting at initial (approximately 2-week) postoperative follow-up
* Prior management of isolated fracture or multi-trauma

Exclusion Criteria:

* Incarceration
* Problems, in the judgement of study personnel, with maintaining follow-up
* Cognitive disability (either acute or chronic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who agree to enroll | 6 months
  Feasibility will be assessed based on percentage of patients who agree to enroll sessions
Score on Modified Treatment Evaluation Inventory Short Form | 6 months
  Acceptability will be measured qualitatively and using the Modified Treatment Evaluation Inventory Short Form
Percentage of patients who complete 5 out of 8 possible Behavioral Activation sessions | 6 months
  Feasibility will be assessed based on patients who complete 5 out of 8 possible Behavioral Activation Sessions

SECONDARY OUTCOMES:
Score on PROMIS general health survey (Response range is 0 to 100 where 100 indicates better function) | 6 months
  Preliminary efficacy on functional outcome will be assessed using patient reported functional outcome using PROMIS general health survey
Score on VAS pain score (Response range is from 0 to 10 where 10 indicates greater pain) | 6 months
  Pain-related preliminary efficacy will be assessed using patient reported VAS pain score will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No